CLINICAL TRIAL: NCT01366430
Title: Treatment of Geotropic Horizontal Canal Benign Paroxysmal Positional Vertigo; Randomized Controlled Trial of Barbeque Rotation and Gufoni Maneuver
Brief Title: Treatment of Geotropic Horizontal Canal Benign Paroxysmal Positional Vertigo
Acronym: HC BPPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chonbuk National University (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: KONOS, Korean neuro-ophthalmology and neuro-otology society
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Treatment of HC BPPV
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2009-01

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: BPPV(benign paroxysmal positional vertigo); HC-BPPV(BPPV involving the horizontal semicircular canal); Nystagmus; Treatment outcome; Horizontal Canal Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Nystagmus, Pathologic | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gefoni manenuver (Active Comparator): Gefoni manenuver for Geotropic HC-BPPV
  Interventions: Procedure: Gufoni
- sham maneuver (Active Comparator): sham maneuver for geotropic HC-BPPV
  Interventions: Procedure: Sham
- barbecue maneuver (Active Comparator): barbecue maneuver for geotropic HC-BPPV
  Interventions: Procedure: Barbecue

INTERVENTIONS:
Procedure: Gufoni — For Gufoni maneuver, the patient was quickly brought down on the healthy side from the sitting position, and the head was then turned about 45 degree down, so that the nose was on the bed. After 2 minutes in this position, the patient was returned to the upright position.
  Arms: Gefoni manenuver
Procedure: Sham — The sham maneuver the opposite of the first step for barbecue rotation; lying down from sitting position for 30 seconds, and head turn 90degree to the affected side for 1 minute, and then sit up.
  Arms: sham maneuver
Procedure: Barbecue — For barbecue rotation, the head was rotated rapidly 90degree while supine in the direction of the healthy ear, which was immediately followed by a truncal rotation of 90degree in the same direction to lie on the intact side. After 30-60 seconds when the induced nystagmus was dissipated, the patients were subjected to a further 90degree rotation of the head and trunk en block in the same direction to attain the nose-down position. After a further 30-60 seconds, the head was again turned in the same direction so that the affected ear was downward. Finally, after another 30-60s, the patient was brought to sitting position. Only one maneuver was performed per session.
  Arms: barbecue maneuver

SUMMARY:
The purpose of this study was to compare the immediate efficacies of each treatment maneuvers in treatment of geotorpic horizontal canal benign paroxysmal positional vertigo (HC-BPPV).

DETAILED DESCRIPTION:
A randomized prospective study of patients with HC-BPPV. Patients with geotropic type of HC-BPPV were randomized to one of each three treatment groups at their first clinic visit. These groups included the barbecue maneuver, Gufoni's maneuver, and sham group in geotropic HC-BPPV. Responsiveness of treatment maneuver was determined by positioning maneuver immediately after each treatment method based on resolves of vertigo and positional nystagmus.

ELIGIBILITY:
Inclusion Criteria:

* a history of brief episodes of positional vertigo, direction-changing horizontal nystagmus beating toward the uppermost (apogeotropic nystagmus) ear in both the lateral head turning positions,
* no spontaneous nystagmus during upright sitting position
* absence of identifiable central nervous system disorders that could explain the positional vertigo and nystagmus

Exclusion Criteria:

* central positional nystagmus with identifiable CNS lesions that could explain the positional nystagmus

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Immediate therapeutic effects for the treatment of geotropic HC-BPPV | one hour
  The immediate treatment response was determined by participating neurologists in each clinic without knowing the maneuver applied to each patient from 30 minutes to one hour after initial maneuver. The absence of both vertigo and nystagmus was required to determine a resolution. When the patient still showed positioning nystagmus or vertigo, the patient received the previously applied maneuver again.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Chonbuk National University Hospital, Jeonju, Cholabuk-do
  - Chonnam National University Hospital, Kwangju, Cholanam-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do